CLINICAL TRIAL: NCT06989099
Title: Lymphedema Prevention Through Immediate Lymphatic Reconstruction (LILY) Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-0255; NCI-2024-05054 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-05-09; First posted 2025-05-25 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Postoperative Evaluations (Experimental): Participants who agree to take part in this study, clinic visit timing will be exactly the same time as would ordinarily be scheduled: before surgery, then 6, 12, 18, and 24 months after surgery. Each study visit should take about 2-3 hours.
  Interventions: Procedure: Immediate Lymphatic Reconstruction (ILR)/; Procedure: Prophylactic Lymphovenous Bypass (pLVB)

INTERVENTIONS:
Procedure: Immediate Lymphatic Reconstruction (ILR)/ — Given by Procedure
Procedure: Prophylactic Lymphovenous Bypass (pLVB) — Given by Procedure

SUMMARY:
To learn if reconstruction of the lymphatic system at the time of axillary lymphadenectomy can reduce the risk of developing lymphedema.

DETAILED DESCRIPTION:
Primary Objectives

- To determine the freedom from lymphedema (FFL) rate at 2 years postoperatively in participants with a diagnosis of IBC undergoing ILR at the time of ALND.

Secondary Objectives

* Estimate the proportion of participants who have lymphedema that persists at 2 years after ILR surgeries.
* Determine baseline lymphatic vessel anatomical or functional characteristics associated with increased risk of lymphedema following ILR.
* Evaluate changes in systemic inflammatory mediators and systemic immune cell function affiliated with lymphedema development.

ELIGIBILITY:
Inclusion Criteria:

1. Participants diagnosed with IBC.
2. Participants who have been scheduled for ILR/pLVB by their treating physician/surgeon at the time of their axillary lymphadenectomy for breast cancer
3. Participants willing and able to comply with the study protocol requirements and all study-related visit requirements.
4. Female subjects at least 18 years old and capable of providing consent to participate.
5. Females of childbearing potential must have a negative urine pregnancy test within 36 hours prior to study drug administration and agree to use a medically accepted method of contraception for a period of one month following the study.

Exclusion Criteria:

1. Patients known to be pregnant or breast-feeding.
2. Patients with known or suspected iodine or ICG hypersensitivity.
3. Patients unable to remain stationary for one hour.
4. Active cellulitis.
5. Subjects with a preoperative clinical lymphedema diagnosis.
6. Subjects undergoing bilateral ALND.
7. Subjects requiring immediate chest wall reconstruction with a pedicled or microvascular flap, or those that have received preoperative radiation therapy.
8. Patients with BMI >45kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from lymphedema (FFL) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Schaverien, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT06989099/Prot_ICF_000.pdf